CLINICAL TRIAL: NCT03169049
Title: Peripheral Nerve Conduction Block Using a High Frequency Alternating Stimulation: A Pilot Study
Brief Title: Nerve Conduction Block Using Transcutaneous Electrical Currents
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Castilla-La Mancha (Other)
Collaborators: Hospital Nacional de Parapléjicos de Toledo (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: ddsm10
Record Dates: First submitted 2017-05-25; First posted 2017-05-30 (Actual); Last update posted 2017-05-30 (Actual); Status verified 2017-05

CONDITIONS: Nerve Block; Electric Stimulation
Keywords: nerve conduction block; high frequency stimulation; handgrip

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High-Frequency (Experimental): Transcutaneous application of high frequency electrical current over the arm for a 20 minutes session. The intensity of the current will increase until participants report a "strong but comfortable" sensation, just below motor threshold.
  Interventions: Device: High-Frequency Stimulation
- Sham stimulation (Sham Comparator): Electrodes are placed over the arm for a 20 minutes in the same manner as experimental group but will be applied a sham electrical stimulation increasing the current intensity of an unconnected channel
  Interventions: Device: sham Stimulation

INTERVENTIONS:
Device: High-Frequency Stimulation — high-Frequency electrical stimulation over superficial ulnar and median nerve through the electrotherapy device Myomed 932. (Enraf-Nonius, Delft, Netherlands)
  Arms: High-Frequency
Device: sham Stimulation — Sham transcutaneous electrical stimulation over superficial ulnar and median nerve through the electrotherapy device Myomed 932. (Enraf-Nonius, Delft, Netherlands)
  Arms: Sham stimulation

SUMMARY:
The purpose of this study is to determine whether the transcutaneous application of unmodulated high frequency alternating currents could produce a quickly conduction block of peripheral nerve.

DETAILED DESCRIPTION:
In the last years several animal experimental studies have evidenced that high frequency unmodulated currents about 5 KHz can cause a peripheral nerve block. However electric currents with these high frequencies that are usually used for the treatment of pain in humans are interrupted or modulated (i.e. interferential currents).

It has show that the diameter of the nerve it is related with the frequency to produce the conduction block. For this reason the investigators decided to applied 20KHz to observe the effects on maximal manual force and to compare versus sham stimulation.

Only one study has applied 5KHz on experimental pain and they have demonstrated changes in somatosensory thresholds.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers

Exclusion Criteria:

* Neuromuscular disease.
* Epilepsy.
* Trauma, surgery or pain affecting the upper limb, shoulder girdle or cervical area.
* Osteosynthesis material in the upper limb.
* Diabetes.
* Cancer.
* Cardiovascular disease.
* Pacemaker or other implanted electrical device.
* Take any drug (NSAIDs, corticosteroids, antidepressants, analgesics, antiepileptics, ...) during the study and in the previous 7 days.
* Presence of tattoos or other external agent introduced into the treatment or assessment area.
* Pregnancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2017-07 (Estimated); Primary Completion 2017-08 (Estimated); Study Completion 2017-09 (Estimated)

PRIMARY OUTCOMES:
Baseline Hand Muscle Strength | Baseline at 0 min
  The hand muscle strength will be measured with a dynamometer and will be expressed in Newton
Hand muscle strength after treatment 20 min | After treatment 20 min
  The hand muscle strength will be measured with a dynamometer and will be expressed in Newton

SECONDARY OUTCOMES:
Change from baseline in Muscle strength | baseline at 0 min, immediately after treatment at 20 min
  The hand muscle strength will be measured with a dynamometer and will be expressed in Newton

CONTACTS AND LOCATIONS:
Overall Officials: Diego Serrano-Muñoz, MsC, Principal Investigator — Hospital Nacional de Parapléjicos, Toledo

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Serrano-Munoz D, Avendano-Coy J, Simon-Martinez C, Taylor J, Gomez-Soriano J. Effect of high-frequency alternating current transcutaneous stimulation over muscle strength: a controlled pilot study. J Neuroeng Rehabil. 2018 Nov 12;15(1):103. doi: 10.1186/s12984-018-0443-2. PMID 30419966